CLINICAL TRIAL: NCT03402022
Title: Drug Use During a Very Long Distance Mountain Trail: a Study Using Automated Urine Collection
Brief Title: Drug Use and Ultra-endurance Race
Acronym: Ultra-Trail
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.049; 2017-A00484-49 (Other: ID RCB)
Record Dates: First submitted 2017-12-15; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Healthy Individuals
Keywords: Sport; competition; ultra-endurance; trail running; doping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — 466 urine samples have been collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypothesis: To verify whether the use of drugs, in particular performance-enhancing drugs, is prevalent amongst participants in a very long distance mountain trail.

Primary objective : To qualify and quantify drug use amongst participants in a very long distance mountain trail, by targeting the molecules most likely used by the runners.

DETAILED DESCRIPTION:
Introduction : very long distance mountain trail which is particularly demanding for the organism. This kind of competition is likely to have an impact on the athlete's health and / or physical integrity. It is assumed that many participants may use medication in an attempt to i) prevent and /or treat medical conditions induced by prolonged muscular exercise, and ii) delay fatigue and improve physical and/or psychological capacities. Beyond ethical and regulatory considerations, such practice in this isolated environment is not without health risks. However, to our knowledge, there is no objective data on medication use during very long distance mountain trails.

Methodology : Individual urine samples from male competitors participating in a very long distance mountain trail and using temporary urinals near the starting line will be collected within three hours before departure, anonymously, blindly, using hidden automated samplers. Simultaneously with automated urine sampling, demographic data (age class, ranking class, geographical area of residence, performance class over the year) will be collected anonymously via an automated system detecting the runners' electronic bibs. The quantification of different classes of drugs in the urine samples will be performed by World Anti-Doping Agency-accredited laboratories using liquid chromatography, mass spectrometry and / or gas chromatography. The classes of molecules sought will be the following: most common non-steroidal anti-inflammatory drugs (NSAIDs), glucocorticoids, stimulants, narcotics, anabolic agents, metabolic modulators, cannabinoids, beta2-agonists, beta-blockers, diuretics, benzodiazepines. A questionnaire about drug use before/during the race and using the randomized response technique (RRT) will be proposed online, anonymously to female and male participant after the competition.

Expected results : drug use is frequent amongst participants in a very long distance mountain trail. Drug use prevalence measured from automated urine collection is higher than that obtained from the RRT questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Automated urine collection : male participants starting a very long distance mountain trail.
* Questionnaire: female and male participants in a very long distance mountain trail.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 2923 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
To measure urinary drug concentrations (in ng/ml) amongst male participants in a very long distance mountain trail, by targeting the molecules most likely used by the runners. | 18 months
  * sampling 466 individual urine specimens from male participants in a very long distance mountain trail;
  * measuring urinary concentrations of drugs belonging to the following classes : nonsteroidal anti-inflammatory drugs (NSAIDs), glucocorticoids, stimulants, narcotics, anabolic agents, metabolic modulators, cannabinoids, beta2-agonists, beta-blockers, diuretics, benzodiazepines. Drug concentrations will be determined through liquid chromatography, mass spectrometry and / or gas chromatography, according to the molecules.

SECONDARY OUTCOMES:
To measure the responses (yes or no) to a questionnaire about drug use, amongst female and male participants in a very long distance mountain trail, by targeting the molecules most likely used by the runners. | 6 months
  - obtaining a return rate of at least 30% to the anonymous, online questionnaire proposed to the participants after their race.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre BOUZAT, Dr, Principal Investigator — University Hospital, Grenoble
Locations (1):
- UniversityHospitalGrenoble, Grenoble, France

REFERENCES:
- [Background] de Hon O, Kuipers H, van Bottenburg M. Prevalence of doping use in elite sports: a review of numbers and methods. Sports Med. 2015 Jan;45(1):57-69. doi: 10.1007/s40279-014-0247-x. PMID 25169441
- [Background] Dietz P, Ulrich R, Dalaker R, Striegel H, Franke AG, Lieb K, Simon P. Associations between physical and cognitive doping--a cross-sectional study in 2.997 triathletes. PLoS One. 2013 Nov 13;8(11):e78702. doi: 10.1371/journal.pone.0078702. eCollection 2013. PMID 24236038
- [Background] McAnulty S, McAnulty L, Nieman D, Morrow J, Dumke C, Henson D. Effect of NSAID on muscle injury and oxidative stress. Int J Sports Med. 2007 Nov;28(11):909-15. doi: 10.1055/s-2007-964966. Epub 2007 May 31. PMID 17541866
- [Background] Millet GY, Banfi JC, Kerherve H, Morin JB, Vincent L, Estrade C, Geyssant A, Feasson L. Physiological and biological factors associated with a 24 h treadmill ultra-marathon performance. Scand J Med Sci Sports. 2011 Feb;21(1):54-61. doi: 10.1111/j.1600-0838.2009.01001.x. PMID 19883385
- [Background] Robach P, Trebes G, Lasne F, Buisson C, Mechin N, Mazzarino M, de la Torre X, Roustit M, Kerivel P, Botre F, Bouzat P. Drug Use on Mont Blanc: A Study Using Automated Urine Collection. PLoS One. 2016 Jun 2;11(6):e0156786. doi: 10.1371/journal.pone.0156786. eCollection 2016. PMID 27253728
- [Derived] Robach P, Trebes G, Buisson C, Mechin N, Mazzarino M, Garribba F, Roustit M, Quesada JL, Lefevre B, Giardini G, DE Seigneux S, Botre F, Bouzat P. Prevalence of Drug Use in Ultraendurance Athletes. Med Sci Sports Exerc. 2024 May 1;56(5):828-838. doi: 10.1249/MSS.0000000000003374. Epub 2024 Jan 18. PMID 38233983